CLINICAL TRIAL: NCT03876691
Title: The Attendance to SHARE Model Communication Course by Physicians Increases the Signing of Do-not-resuscitate Orders for Critical Patients in the Emergency Room
Brief Title: SHARE Model Communication Course and Do-not-resuscitate Signing
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG8G0681
Record Dates: First submitted 2019-02-25; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries | interventions — Physicians

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Do not resuscitate: Patients who are suggested to family about a do-not-resuscitate order treatment by physicians.
  Interventions: Other: Patients; Other: Physician

INTERVENTIONS:
Other: Patients — Patients who are considered as terminally ill and would not benefit from aggressive treatment, who physicians suggest to family about a do-not-resuscitate.
Other: Physician — The current emergency medical department departments within the preparation of the attending physician

SUMMARY:
This study aimed to investigate the effect of attending a SHARE model communication course by emergency physicians on patient notification and signing of do-not-resuscitate (DNR) orders for critical patients in the emergency room.

DETAILED DESCRIPTION:
An observation form designed based on the SHARE model was completed by two observers who noted the communication process between physicians and patients and family members during patient notification and signing a DNR order. To assess the influence of physicians attending a SHARE model course on the signing of DNR orders, a propensity score-matched population was created to reduce the potential selection bias of patients and family members.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are considered as terminally ill and would not benefit from aggressive treatment, who physicians suggest to family about a "Do not resuscitate" order.
* Patients who was not register with "Do- not- resuscitate" on their health insurance card.

Exclusion Criteria:

* Trauma patients.
* Suicide patients.
* Patients of age less than 20.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research subjects consisted of attending physicians, who were willing to inform consent forms, in the emergency department between May 2017 and April 2018.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with DNR singing observation form | up to 5 months
  The content of the observation form was filled by observers during the explanation process

CONTACTS AND LOCATIONS:
Overall Officials: TSANG-TANG Hsieh, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan